CLINICAL TRIAL: NCT04189952
Title: A Phase 2, Open-Label Study of Acalabrutinib in Combination With R-ICE For Relapsed or Refractory Non-Germinal Center Diffuse Large B Cell Lymphoma, Transformed Chronic Lymphocytic Leukemia/Small Lymphocytic Leukemia or Transformed Marginal Zone Lymphoma
Brief Title: Acalabrutinib in Combination With R-ICE For Relapsed or Refractory Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator Decision
Sponsor: University of Miami (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Craig Moskowitz, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190706
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Results first posted 2022-09-19 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Diffuse Large B Cell Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Leukemia; Marginal Zone Lymphoma
Keywords: Non-Germinal Center Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — acalabrutinib; Rituximab; Ifosfamide; Carboplatin; Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acalabrutinib + R-ICE (Experimental): Acalabrutinib in combination with rituximab, ifosfamide, carboplatin and etoposide (R-ICE). All participants will receive combination treatment for 3 cycles. Each cycle lasts 21 consecutive days. Combination treatment includes twice daily dose of Acalabrutinib, Rituximab on Day 1 of each cycle, Ifosfamide and Carboplatin on Day 2 of each cycle, and Etoposide on Days 1-3 of each cycle.
  Interventions: Drug: Acalabrutinib; Drug: Rituximab; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib 100 mg capsules taken by mouth every 12 hours (PO BID), for a total of 2 daily doses on Days 1 to 21 of each cycle.
  Other Names: ACP-196
Drug: Rituximab — Rituximab 375 mg/m2 administered intravenously (IV) on Day 1 of each cycle.
  Other Names: Rituxan
Drug: Ifosfamide — Ifosfamide 5g/m2 administered intravenously (IV) over 24 hours on Day 2 of each cycle.
  Other Names: Ifex; Isophosphamide
Drug: Carboplatin — Carboplatin Area Under the Concentration time Curve (AUC) 5 IV administered intravenously (IV) on Day 2 of each cycle.
  Other Names: Paraplatin
Drug: Etoposide — Etoposide 100 mg/m2 administered intravenously (IV) on Days 1, 2 and 3 of each cycle.
  Other Names: Etopophos; Toposar; VePesid

SUMMARY:
The purpose of this study is to test a combination treatment of acalabrutunib when given together with rituximab-ifosfamide-carboplatin-etoposide (R-ICE) to evaluate if it will be able to improve durable responses and cure some patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age.
2. Patients must have histologic confirmation of relapsed or refractory lymphoma.
3. Baseline FDG-PET scans must demonstrate positive lesions compatible with CT defined anatomical tumor sites.

   a) CT scan showing at least:
   * i. 2 or more clearly demarcated lesions/nodes with a long axis >1.5cm and short axis ≥ 1.0cm, or
   * ii. 1 clearly demarcated lesion/node with a long axis >2.0cm and short axis ≥1.0cm.
4. Patient must have been previously treated for B cell non-Hodgkin lymphoma with any of the allowable below:

   1. First-line treatment with rituximab and an anthracycline-based chemotherapy.
   2. Monotherapy rituximab, dosed prior to first-line rituximab combined with anthracycline containing chemotherapy, or as maintenance therapy.
   3. Radiotherapy as part of the first-line treatment plan including anthracycline and rituximab.
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
6. Life expectancy of greater than 6 weeks.
7. Patients must have normal organ and marrow function as defined below,

   1. absolute neutrophil count ≥ 1000/microliters (mcL) (unless due to lymphoma involvement of the bone marrow),
   2. platelets ≥75,000/mcL (unless due to lymphoma involvement of the bone marrow),
   3. total bilirubin <1.5 x within normal institutional limits (unless due to lymphoma involvement of liver or a known history of Gilbert's disease),
   4. Aspartate transaminase (AST) (SGOT)/Alanine transaminase (ALT) (SGPT) ≤ 2.5 × institutional upper limit of normal (unless due to lymphoma involvement of liver),
   5. creatinine within normal institutional limits, or
   6. creatinine clearance ≥40 mL/min/1.73 m2 for patients with creatinine levels above institutional normal. (unless due to lymphoma).
8. Major surgical procedure within 28 days of first dose of study drug. If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
9. Women who are sexually active and can bear children must agree to use highly effective forms of contraception during the study and for 90 days after the last dose of acalabrutinib + R-ICE.
10. Men who are sexually active and can beget children must agree to use highly effective forms of contraception during the study and for 90 days after the last dose of acalabrutinib + R-ICE.
11. Men must agree to refrain from sperm donation during the study and for 90 days after the last dose of study drug.
12. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty.
13. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations).

Exclusion Criteria:

1. Germinal-center cell-of-origin DLBCL.
2. Patients who have had chemotherapy or radiotherapy < 21 days prior to first administration of study treatment or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
3. Patients who are receiving any other investigational agents.
4. Patients with known central nervous system involvement of lymphoma.
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to acalabrutinib or R-ICE with the exception of first-infusion reaction to rituximab.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Recent infections requiring systemic treatment need to have completed therapy > 7 days before the first dose of study drug.
7. Pregnant women are excluded from this study because an acalabrutinib R-ICE is a chemotherapy program with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with acalabrutinib R-ICE, breastfeeding should be discontinued if the mother is treated with acalabrutinib R-ICE.
8. HIV-positive patients on combination antiretroviral therapy are eligible, unless the patient's CD4 count is below the institutional lower limit of normal, or the patient is taking prohibited CYP3A4/5 strong inhibitors or inducers.
9. Patients may not have received any anti-cancer therapy for their primary rel/ref DLBCL with the exception of palliative radiation therapy (RT).
10. Uncontrolled Autoimmune Hemolytic Anemia or immune thrombocytopenia purpura (ITP) resulting in (or as evidenced by) declining platelet or Hgb levels within the 4 weeks prior to first dose of study drug.
11. Presence of transfusion-dependent thrombocytopenia.
12. Prior exposure to a Bruton's tyrosine kinase (BTK) inhibitor.
13. History of prior malignancy, with the exception of the following:

    1. Malignancy treated with curative intent felt to be at low risk for recurrence by treating physician,
    2. Adequately treated non-melanomatous skin cancer or lentigo maligna melanoma without current evidence of disease,
    3. Adequately treated cervical carcinoma in situ without current evidence of disease.
14. Currently active clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure, or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification, or history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to first dose with study drug.
15. Unable to swallow capsules, or disease significantly affecting gastrointestinal function or, resection of the stomach or small bowel, or symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
16. Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody will need a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive patients will be excluded.) Hepatitis C antibody positive patients are eligible if PCR is negative. Hepatitis B core antibody (+) patients without evidence of HBsAg or Hep B PCR (+) are eligible with appropriate Hepatitis B reactivation prophylaxis.
17. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
18. Current life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the patient's safety, or put the study at risk.
19. Received anticoagulation therapy with Coumadin or equivalent vitamin K antagonists within the last 28 days.
20. Vaccinated with live, attenuated vaccines with 4 weeks of first does of study drug.
21. Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 5), grade ≤1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia.
22. Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia.
23. Unwilling or unable to participate in all required study evaluations and procedures.
24. Currently active, clinically significant hepatic impairment (≥ moderate hepatic impairment according to the NCI/Child Pugh classification.
25. Breastfeeding or pregnant.
26. Concurrent participation in another therapeutic clinical trial.
27. Patients who require proton pump inhibitors at baseline (prior to fist dose of study drug) or strong CYP3A4 inhibitor or inducer and are not able to switch to another medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Moskowitz, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period
Arm/Group | Acalabrutinib + R-ICE
Started | 2
Completed | 2
Not Completed | 0
Period: Follow-up Period
Arm/Group | Acalabrutinib + R-ICE
Started | 2
Completed | 0
Not Completed | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Acalabrutinib + R-ICE
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Complete Response (CR)
Description: The percentage of participants achieving complete response (CR) will be assessed using Response Evaluation Criteria in Lymphoma (RECIL 2017) criteria.
Time Frame: 9 weeks (End of Cycle 3)
Measure: Number; unit: percentage of participants
Arm/Group | Acalabrutinib + R-ICE
Number analyzed (Participants) | 2
percentage of participants | NA — Results not reported due to participant confidentiality.

2. Secondary Outcome: Number of Treatment-Emergent Adverse Events
Description: The safety profile and tolerability of acalabrutinib + R-ICE will be reported as the number of treatment-emergent adverse events (AEs) or abnormalities of laboratory tests; serious adverse events (SAEs); dose-limiting toxicities (DLTs), or AEs leading to discontinuation of study treatment, or death. Severity and relationship will be assessed by the treating physician using the Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.
Time Frame: 13 weeks
Measure: Number; unit: Treatment-emergent adverse events
Arm/Group | Acalabrutinib + R-ICE
Number analyzed (Participants) | 2
Treatment-emergent adverse events | NA — Results not reported due to participant confidentiality.

3. Secondary Outcome: Percentage of Participants Achieving Partial Response (PR)
Description: The percentage of participants achieving partial response (PR) will be assessed using Response Evaluation Criteria in Lymphoma (RECIL 2017) criteria.
Time Frame: 9 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Acalabrutinib + R-ICE
Number analyzed (Participants) | 2
percentage of participants | NA — Results not reported due to participant confidentiality.

4. Secondary Outcome: Percentage of Participants Achieving Overall Response
Description: Overall response is defined as the percentage of participants who achieved complete response (CR) or partial response (PR) to acalabrutinib + R-ICE therapy. Response will be assessed using Response Evaluation Criteria in Lymphoma (RECIL 2017) criteria.
Time Frame: 9 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Acalabrutinib + R-ICE
Number analyzed (Participants) | 2
percentage of participants | NA — Results not reported due to participant confidentiality.

5. Secondary Outcome: Percentage of Participants Achieving Mobilization Rate Greater Than or Equal to 2x10^6 CD34+ Cells/kg Body Weight
Description: Percentage of study participants achieving a mobilization rate of greater than or equal to 2x10^6 CD34+ cells/kg body weight. Descriptive statistics will be used to summarize the mobilization rates.
Time Frame: 9 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Acalabrutinib + R-ICE
Number analyzed (Participants) | 2
percentage of participants | NA — Results not reported due to participant confidentiality.

6. Secondary Outcome: Event-Free Survival (EFS)
Description: Duration of Event-Free Survival (EFS) in study participants. EFS is defined as the time from first dose to documented disease progression, death from any cause, or study dropout, whichever occurs first.
Time Frame: Up to 61 weeks
Measure: Number; unit: weeks
Arm/Group | Acalabrutinib + R-ICE
Number analyzed (Participants) | 2
weeks | NA — Results not reported due to participant confidentiality.

7. Secondary Outcome: Progression-Free Survival (PFS)
Description: Duration of Progression-Free Survival (PFS) in study participants. PFS is defined as the time from first dose to documented disease progression, or death from any cause, whichever occurs first. Data for subjects who are still alive and free from progression at the time of data cutoff date, lost to follow-up, or have discontinued the study will be censored on last assessment (or, if no post-baseline tumor assessment, at the time of first dose plus 1 day).
Time Frame: Up to 61 weeks
Measure: Number; unit: weeks
Arm/Group | Acalabrutinib + R-ICE
Number analyzed (Participants) | 2
weeks | NA — Results not reported due to participant confidentiality.

8. Secondary Outcome: Overall Survival (OS)
Description: Duration of Overall Survival (OS) in study participants. OS is defined as the time from first dose to death from any cause. Data for subjects who are still alive at the time of data cutoff date, lost to follow-up, have discontinued the study (or, if no post-baseline assessment, at the time of first dose plus 1 day) will be censored.
Time Frame: Up to 61 weeks
Measure: Number; unit: weeks
Arm/Group | Acalabrutinib + R-ICE
Number analyzed (Participants) | 2
weeks | NA — Results not reported due to participant confidentiality.

ADVERSE EVENTS:
Time Frame: 10 months
Description: Adverse Events not reported due to participant confidentiality.
Arm/Group | Acalabrutinib + R-ICE
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
To protect participant privacy and maintain confidentiality, results will not be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT04189952/Prot_SAP_000.pdf